CLINICAL TRIAL: NCT03989726
Title: Efficacy of High Density Voltage and Fractionation Map Guided Ablation Compared to Anatomy-based Circumferential Pulmonary Vein Isolation in Patients With Atrial Fibrillation
Brief Title: Efficacy of High Density Voltage and Fractionation Map Guided Ablation in Patients With Atrial Fibrillation
Acronym: INVENTION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Keimyung University Dongsan Medical Center (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSMCEP_PHS_003
Record Dates: First submitted 2019-06-14; First posted 2019-06-18 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-06

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High density voltage and fractionation map guided group (Experimental): * Complex fractionated atrial electrogram (CFAE), voltage and fractionation map will be performed with a multielectrode mapping catheter.
  * The mapping should be performed in AF.
  * First, low-voltage zone is defined as an area with bipolar peak-to-peak voltage amplitudes < 0.5mV.
  * A voltage-map guided segmental PV isolation is performed. Radiofrequency energy is applied in the antral regions of the PVs. High voltage zone over 0.5mV in the antral region is targeted. IF PV isolation in not achieved by voltage-guided segmental ablation, additional Lasso catheter guided segmental antral ablation is performed.
  * Radiofrequency energy is delivered at target sites for 15-30 sec guided by contact force, lesion size index (LSI) and local electrogram elimination.
  * If the patient is still in AF after PV isolation, additional fractionation map guided ablation is performed. The fractionation area within low voltage area (<0.5mV) should be targeted.
  Interventions: Procedure: AF ablation
- Circumferential PV isolation (Active Comparator): A control group will be chosen from database of patients who underwent AF ablation between 2018-2019. A control group includes the same number of consecutive patients who underwent anatomy-based circumferential PV isolation.
  Interventions: Procedure: AF ablation

INTERVENTIONS:
Procedure: AF ablation — AF ablation includes pulmonary vein isolation and/or voltage and fractionation guided ablation

SUMMARY:
The purpose of this study is to evaluate the efficacy of high density voltage and fractionation map guided ablation compared to anatomy-based circumferential pulmonary vein Isolation in patients with atrial fibrillation

DETAILED DESCRIPTION:
In this study, a test group includes those who undergoing atrial fibrillation(AF) ablation guided by high density voltage and fractionation map. A control group will be chosen from database of patients who underwent AF ablation between 2018-2019. A control group includes the same number of consecutive patients who underwent anatomy-based circumferential pulmonary vein (PV) isolation.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age over 20 years old and under 80 years old 2. Patients with non-valvular atrial fibrillation 3. Patients having AF even after receiving continued treatment with at least 1 antiarrhythmic drug for more than 6 weeks 4. Patients who can understand the information sheet and consent form on the need and procedure of catheter ablation and submitted them 5. Patients who are available of follow-up at least for more than three months after catheter ablation

Exclusion Criteria:

1. Patients unsuitable for catheter ablation because the size of left atrium is over 6.0 cm
2. Patients unsuitable for catheter ablation due to previous history of pulmonary surgery or structural heat disease.
3. Patients who cannot receive standard treatments such as anticoagulation therapy which need to be continuously performed prior to radiofrequency catheter ablation
4. Patients in the subject group vulnerable to clinical study
5. Patients who had undergone a prior catheter ablation for atrial fibrillation

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Free from atrial arrhythmia at 12 months | 12 months
  Freedom from any atrial arrhythmia lasting longer than 30 seconds during 1 year follow-up after single ablation with or without the use of antiarrhythmic medications with the exclusion of the 3-month blanking period.

SECONDARY OUTCOMES:
Acute AF termination rate during the procedure | During the procedure
  Acute AF termination rate during the procedure
Complication rate | 12 months
  Compare complication rate between two groups
Total procedure time, ablation time, fluoroscopy time | 12 months
  Total procedure time, ablation time, fluoroscopy time between two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Keimyung University Dongsan Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No